CLINICAL TRIAL: NCT04722289
Title: The Together on Diabetes Intervention
Brief Title: The Together on Diabetes Intervention - a Realist Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Diabetes, Copenhagen Municipality (Other Government)
Collaborators: Novo Nordisk A/S (Industry); Innovation Fund Denmark (Individual); University of Copenhagen (Other); The Danish Diabetes Association (Other)
Responsible Party: Principal Investigator, Stine Garn, Evaluator, PhD, Center for Diabetes, Copenhagen Municipality
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDiabetesCopenhagen
Record Dates: First submitted 2021-01-08; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Type 2 Diabetes Mellitus; Health Behavior; Delivery of Health Care
Keywords: Realist evaluation; Complex intervention; Implementation; Mechanism; Contextual factors; Peer support; Health inequalites; Diabetes self-management; Healthcare services
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Health Behavior

STUDY DESIGN:
Intervention Model Description: A multi-method case study approach was used to identify mechanisms generating improved diabetes self-management and use of healthcare services (outcome) Thus, using this method, it enabled to investigate similarities and differences in how the mechanisms operated depending on peers' context.
  All peers and peer supporters included and matched in the intervention from February 2018 to July 2019 were invited by the project manager to participate in this study. In total, 9 out of 12 pairs who completed the intervention during this period accepted the invitation, and were thereby selected as cases. The peers were recruited through CfD (N=7), their GP (N=1), and the home care (N=2). The peer supporters were recruited among people who had completed a patient education in CFD (N=5), by members from the DDA (N=2), their GP (N=1), or by people who applied via 'Together on Diabetes' webpage (N=2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Together on Diabetes (Experimental): The intervention consists of five components: Recruitment of peers and peer supporters; training of peer supporters; matching peers and peer supporters; individual face-to-face meetings between peers and peer supporters; and ongoing supervision and network meetings for peer supporters.
  Interventions: Behavioral: Together on Diabetes

INTERVENTIONS:
Behavioral: Together on Diabetes — Social and emotional support'; 'Assistance in daily management'; and 'Linkage to healthcare services'

SUMMARY:
The Danish healthcare system is universal and free of charge for Danish citizens, as all healthcare services are financed by general taxes. However, socioeconomic differences exist in access to healthcare services, treatment, and consequences of type 2-diabetes (T2D).

Using a realistic evaluation approach, this study aimed to evaluate the implementation of a Danish peer support intervention, targeted on improving self-management and use of healthcare services among socially vulnerable people with type 2-diabetes ("peers"). The study focused on the mechanisms generating the intended outcomes. Further, how contextual factors in peers' everyday life facilitated or hindered the mechanisms to operate.

The study design is a multi-method case study (n=9). Data include qualitative semi-structured interviews with four key groups of informants (peer, peer supporter, project manager, and a diabetes nurse). Each type of informant per case was interviewed (n=25) to obtain different perspectives of how the peers' interacted, and benefited from the intervention. All interviews were completed immediately after the after the 6-month intervention.

Further, a quantitative survey was conducted among peers at baseline (N=9) and follow-up (N=9) to obtain information about how peers' individual contextual factors, such as their sociodemographic characteristics, co-morbidity, diabetes complications, social relations, and other life events influenced how they perceived and interacted in the intervention. Further, to measure improvements in their diabetes-self management (DSM) and use of healthcare services (outcomes). Questions from the Danish National Health Survey were used to measure DSM: (eating habits, physical activity,and medication intake). Use of healthcare services was measured by the number of times (during a 12-month period) the peers' attended diabetes controls at the GP; food therapist, and ophthalmologist or had other form of contacts with relevant health care services.

All data were collected between February 2018 and April 2020.

Hypothesis: 6-month individual face-to-face peer support provided by non-professional persons with T2D can improve self-management and use of healthcare services among socially vulnerable people with T2D if contextual factors such as peers' sociodemographic characteristics, health condition, and social relations facilitate their engagement in the intervention. Potential mechanisms that generate the expected outcomes might be: peers' motivation, trust, perceived beliefs and needs; and experience of being supported by the peer supporters.

DETAILED DESCRIPTION:
The intervention consists of five components: Recruitment of peers and peer supporters; training of peer supporters; match making of peers and peer supporters; individual face-to-face meetings between peers and peer supporters; and ongoing supervision and network meetings for peer supporters. The peer support meetings are held approximately every second week for six months and contain three activities: 'Social and emotional support'; 'Assistance in daily management'; and 'Linkage to healthcare services'

ELIGIBILITY:
Peers:

Inclusion Criteria:

* Poorly regulated T2D
* multi-morbidity
* no employment
* low/no education
* no contact to the healthcare system
* living alone with no/spare social network.

Exclusion Criteria:

- Poor regulated mental disease.

Peer supporters

Inclusion criteria:

* Well-regulated T2D
* Basic knowledge about T2D and the Danish healthcare system;
* Good communication skills
* Empathy
* An interest in supporting a socially vulnerable person with T2D
* Available two hours every second week for at least six-month (the intervention period).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Baseline, diet habits | Assessed among peers before study participation, 0 month
  Peers' diet habits (self-reported), Questionnaire data
Change from Baseline, diet habits at 6 month | Assessed among peers after study participation, at 6 month
  Improvements in the peers' diet habits (self-reported), Questionnaire data
Baseline, physical activity (training) | Assessed among peers before study participation, 0 month
  Peers' physical activity level measured by time spend in a typical week on physiclal acitivty were they are breathing (eg. running, exercise gymnastics or ball sports) (self-reported), Questionnaire data
Change from Baseline, physical activity (training) at 6 month | Assessed among peers after study participation, at 6 month
  Improvements in the peers' physical activity level measured by time spend in a typical week on physiclal acitivty were they are breathing (eg. running, exercise gymnastics or ball sports) (self-reported), Questionnaire data
Baseline, physical activity (everyday activities) | Assessed among peers before study participation, 0 month
  Peers' physical activity level measured by time spend in a typical week on everyday activities (eg. walking, cycling or gardening? (self-reported), Questionnaire data
Change from Baseline, physical activity (everyday activities) at 6 month | Assessed among peers after study participation, at 6 month
  Improvements in the peers' physical activity level measured by time spend in a typical week on everyday activities (eg. walking, cycling or gardening? (self-reported), Questionnaire data
Baseline, diabetes medication adherence | Assessed among peers before study participation, at 0 month
  Peers' diabetes medication adherence measured by how often they forget to take their prescribed diabetes medication (self-reported), Questionnaire data
Baseline, diabetes medication adherence | Assessed among peers before study participation, at 0 month
  Improvements in peers' diabetes medication adherence measured by how often they forget to take their prescribed diabetes medication (self-reported), Questionnaire data
Baseline, Use of healthcare services (diabetes controls at the GP) | ssessed among peers before study participation, 0 month
  Number of diabetes controls at GP (self-reported), Questionnaire data
Change from baseline, use of healthcare services (diabetes controls at the GP) | Assessed among peers after study participation, at 6 month
  Improvements in the number of diabetes controls at the GP (self-reported), Questionnaire data
Baseline, use of healthcare services (diabetes controls at the foot therapist) | Assessed among peers before study participation, at 0 month
  Number of diabetes controls at the food therapist) (self-reported), Questionnaire data
Change from baseline, use of healthcare services (diabetes controls at the foot therapist) | Assessed among peers after study participation, at 6 month
  Improvements in the number of diabetes controls at the food therapist) (self-reported), Questionnaire data
Baseline, use of healthcare services (diabetes controls at the ophthalmologist ) | Assessed among peers before study participation, at 0 month
  Number of diabetes controls at the ophthalmologist ) (self-reported), Questionnaire data
Change from baseline, use of healthcare services (diabetes controls at the ophthalmologist ) | Assessed among peers after study participation, at 6 month
  Improvements in the number of diabetes controls at the ophthalmologist ) (self-reported), Questionnaire data

REFERENCES:
- [Derived] Garn SD, Glumer C, Villadsen SF, Malling GMH, Christensen U. Understanding the mechanisms generating outcomes in a Danish peer support intervention for socially vulnerable people with type 2-diabetes: a realist evaluation. Arch Public Health. 2021 Sep 6;79(1):160. doi: 10.1186/s13690-021-00676-3. PMID 34488884